CLINICAL TRIAL: NCT02012413
Title: Effect of Pulsed Signal Therapy in Patella Chondromalacia. Randomized Prospective Trial.
Brief Title: Effect of Pulsed Signal Therapy in Patella Chondromalacia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marco Kawamura Demange, Assistant Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/50167-6
Record Dates: First submitted 2013-08-08; First posted 2013-12-16 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Patella Chondromalacia
Keywords: knee; chondromalacia; patella; pulsed signal therapy; PST
MeSH Terms: conditions — Chondromalacia Patellae; Cartilage Diseases; Patella Fracture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PST group (Active Comparator): roughly 20 patients will be treated with PST protocol, outcomes will be Kujala score improvement at 3, 6 and 12 months.
  Interventions: Device: PST - Pulsed Signal Therapy
- Control group (Placebo Comparator): roughly 20 patients will be submitted to a placebo PST protocol, outcomes will be Kujala score improvement at 3, 6 and 12 months.
  Interventions: Device: Placebo - Sham PST

INTERVENTIONS:
Device: PST - Pulsed Signal Therapy — PST application is a painless over-the-skin eletromagnetic field application. 9 sessions of application of electromagnetic therapy - PST - during 60 minutes
  Other Names: PST; PEMF; Pulsed Eletromagnetic Field
  Arms: PST group
Device: Placebo - Sham PST — Placebo PST will be performed by applying the same device over the patient knee. The machine is not applying the PST but it appears to be on. In this way, patients are blinded to the intervation.
  9 sessions of application of Sham PST - during 60 minutes
  Other Names: Placebo
  Arms: Control group

SUMMARY:
PST (pulsed signal therapy) is a unique form of pulsed electromagnetic field therapy (PEMF) for stimulating healing of damaged structures such as cartilage, bones and soft tissues. The physical effect of the pulsed electromagnetic field (PEMF) has been focus of research in various studies, with cartilage being the most studied, and which has demonstrated an increase in the synthesis of proteoglican and collagen in vitro. This is an randomized, controlled and double blind clinical trial. The main objective is to evaluate clinical improvement regarding anterior knee pain after PST intervention in patients with patellar condropathy.

DETAILED DESCRIPTION:
The study was approved by the Research Ethics Committee of the Clinical Hospital (Hospital das Clinicas), University of São Paulo (Universidade de São Paulo - USP) under number 0253/11.

This patient population is estimated to a total of 40 knees, with the patients meeting the following inclusion criteria:

* aged between 20 and 50 years;
* male or female;
* patellofemoral pain syndrome without tibiofemoral and trochlear chondral degeneration according to magnetic resonance imaging (MRI);
* presence of patellar chondropathy confirmed by MRI;
* not having started using direct action drugs on the cartilage in the last 6 months;
* absence of prior surgery on the studied knee;
* absence of invasive procedures, such as knee infiltration, in the previous 12 months;
* absence of disease in the contralateral limb that would cause an excessive burden on the studied limb; and
* absence of contraindications to performing PST, including a pacemaker, cancer, infectious disease activity, severe heart failure, arrhythmias, angina, epilepsy and pregnancy.

The presence of patellofemoral pain is identified by anamnesis and physical examination performed by knee surgeons with more than 10 years' experience. The presence of all of the following criteria is required for diagnosis: typical complaint of anterior knee pain with a duration longer than 3 months (when going up or down stairs, squatting, remaining for long periods with bent knees), pain on palpation of the patellar articular surface and pain on patellar compression (reproducing the patient's complaint).

After inclusion in the study, all of the patients will be instructed (for the duration of the study) not to use drugs with a direct action on the cartilage (e.g., chondroprotectors, such as glucosamine and chondroitin) to avoid confounding biases regarding the effects of the treatments. No patients will be included who had started using these drugs in the previous 6 months to avoid the initial effect of this treatment being a confounder in terms of clinical improvement.

The study is designed so that the patient and the orthopedist evaluating the clinical outcome do not know to which group the patient belongs (i.e., a double-blind study).

After patient inclusion and signing of the terms of free and informed consent, the patients will be randomized by a computer into 2 equal groups, i.e., the control and PST groups. The patients with both knees included in the study will receive randomization for the right knee, and the left will be automatically allocated into the other group. This method was selected to best demonstrate any differences between groups. The final distribution of patients into groups will be therefore not equalized.

PST application will be then directed to the patellofemoral joint. The PST application protocol is as follows: 9 daily 1-hour applications, with 5 in the first week, a break for the weekend, and 4 more the following week.

The control group patients will be submitted to placebo PST treatment with the same protocol and the device connected not generating magnetic pulses. The device operates silently, and it is not possible for the patient to determine whether they are receiving the placebo or treatment, thus maintaining patient blinding. For patients with both knees included, 9 sessions of the treatment are performed on one side and 9 more sessions of the placebo on the other.

All of the participants are instructed to maintain their usual level of physical activity.

The Kujala score will be taken after 3, 6 and 12 months in both groups. If superiority of the PST group is observed, it was decided for ethical reasons that the placebo group should receive the PST treatment and would again be followed up for 1-year post-treatment, with the Kujala score ascertained at 3, 6 and 12 months.

A sample of approximately 20 patients in each group was used for an alpha of 5% and beta of 20%. An effect size of 8 to 10 between groups was sought and is considered clinically significant in terms of Kujala score.

ELIGIBILITY:
Inclusion Criteria:

* patellofemoral pain syndrome without tibiofemoral and trochlear chondral degeneration according to magnetic resonance imaging (MRI);
* presence of patellar chondropathy confirmed by MRI;
* not having started using direct action drugs on the cartilage in the last 6 months;
* absence of prior surgery on the studied knee;
* absence of invasive procedures, such as knee infiltration, in the previous 12 months;
* absence of disease in the contralateral limb that would cause an excessive burden on the studied limb; and
* absence of contraindications to performing PST, including a pacemaker, cancer, infectious disease activity, severe heart failure, arrhythmias, angina, epilepsy and pregnancy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical improvement - Kujala score | 12 months
  A functional score (Kujala) will be performed before, at 3 months, at 6 months and at one year after PST intervention and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Lucia P Silva, B.Sc., M.Sc., Principal Investigator — University of Sao Paulo; Riccardo G Gobbi, M.D., Principal Investigator — University of Sao Paulo; Gilberto L Camanho, M.D., Ph.D, Study Chair — University of Sao Paulo; Marco K Demange, M.D., Ph.D, Study Director — University of Sao Paulo
Locations (1):
- Hospital das Clínicas - Universty of São Paulo, São Paulo, Brazil